CLINICAL TRIAL: NCT01785745
Title: Evaluation of the Effectiveness of Neurocognitive Therapeutic Exercise in Pain Control and Functional Recovery of the Shoulder Impingement Syndrome in Comparison With Traditional Therapeutic Exercise
Brief Title: Study of Neurocognitive Therapeutic Exercise in the Shoulder Impingement Syndrome in Comparison With Traditional Therapeutic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Bertolini, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 486/2012
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Shoulder Impingement Syndrome
Keywords: conservative treatment; shoulder; neurocognitive therapeutic exercise; traditional therapeutic exercise; pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional therapeutic exercise (Active Comparator): The traditional exercise protocol contains mainly strengthening exercises, stretching exercises, Codman's pendulum exercises and exercises against elastic band resistance.
  Interventions: Other: Traditional therapeutic exercise
- Neurocognitive therapeutic exercise (Experimental): The neurocognitive exercise protocol contains ten exercises involving specific instruments (e.g., table inclined with a board with five concentric circles, sponges of various texture).
  Interventions: Other: Neurocognitive therapeutic exercise

INTERVENTIONS:
Other: Neurocognitive therapeutic exercise — Ten exercises involving specific instruments (e.g., table inclined with a board with five concentric circles, sponges of various texture). One-hour session for three times a week for five weeks.
  Arms: Neurocognitive therapeutic exercise
Other: Traditional therapeutic exercise — Different exercises as strengthening exercises, stretching exercises, Codman's pendulum exercises and exercises against elastic band resistance. One-hour session for three times a week for five weeks
  Arms: Traditional therapeutic exercise

SUMMARY:
It is a single-blind randomized controlled clinical trial to evaluate the effectiveness of neurocognitive therapeutic exercise in subjects affected by shoulder impingement syndrome in comparison with traditional therapeutic exercise. The traditional exercise protocol contains mainly strengthening exercises, stretching exercises, Codman's pendulum exercises and exercises against elastic band resistance. The neurocognitive exercise protocol contains ten exercises involving specific instruments (e.g., table inclined with a board with five concentric circles, sponges of various texture). Each subject, randomly assigned to either neurocognitive therapeutic exercise (group 1) or traditional therapeutic exercise (group 2), will be submitted to one-hour session for three times a week for five weeks. The outcome measures used will be the Quick-DASH questionnaire, the Constant-Murley shoulder outcome score, the ASES score, a visual analogic scale (VAS) and the assessment will be performed at baseline (T0), at the end of treatment protocol (T1), at 3 months (T2) and 6 months (T3) from the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with shoulder impingement syndrome established by clinical examination, X-ray in anteroposterior, axillary and outlet views, and magnetic resonance imaging (MRI) or echography.

Exclusion Criteria:

* Rotator cuff and/or subscapularis tendon partial/full-thickness tears,
* capsulolabral pathology responsive to surgical repair,
* congenital abnormalities of the acromion,
* previous surgery on the affected shoulder,
* inflammatory or neurological (systemic or local) diseases involving shoulder girdles,
* cognitive or psychiatric disorders,
* local tumor metastasis or application of radiotherapy,
* acute infections or osseous tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
changing of the Quick-DASH, the short form of the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | baseline (T0), five weeks (T1), three months (T2), six months (T3)
  Assessment of changing of the physical ability and symptoms of the upper extremity

SECONDARY OUTCOMES:
changing of the Constant-Murley shoulder outcome score | baseline (T0), five weeks (T1), three months (T2), six months (T3)
  assessment of changing in shoulder range of motion, pain and strength
changing of the American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form (ASES) score | baseline (T0), five weeks (T1), three months (T2), six months (T3)
  Assessment of changing of the physical ability on daily-living tasks
changing of the visual analogic scale (VAS) | baseline (T0), five weeks (T1), three months (T2), six months (T3)
  assessment of changing of shoulder Pain at rest
changing of the visual analogic scale (VAS) | baseline (T0), five weeks (T1), three months (T2), six months (T3)
  assessment of changing of shoulder Pain during movements
changing of the Likert score | baseline (T0), five weeks (T1), three months (T2), six months (T3)
  assessment of changing in participant satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital "A. Gemelli", Catholic University of the Sacred Heart, Rome, Italy, Italy